CLINICAL TRIAL: NCT04869501
Title: Expanded Access Protocol for an Intermediate Size Population-use of TJ004309 in Combination With Atezolizumab (Tecentriq®) in Patients With Advanced or Metastatic Cancer
Brief Title: Expanded Access Study of TJ004309 in Patients With Advanced or Metastatic Cancer
Status: No longer available | Type: Expanded Access
Sponsor: I-Mab Biopharma US Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: TJ004309STM104
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: TJ004309 — Antibody to CD73
Drug: Atezolizumab — Humanized monoclonal antibody to PD-L1
  Other Names: Tecentriq

SUMMARY:
This expanded access protocol was designed to provide TJ004309 in combination with atezolizumab to the remaining three patients with advanced or metastatic cancer who plan to continue with treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in the Tracon sponsored 4309ST101 or I-Mab sponsored TJ004309STM103 study and thought to have potential to derive clinical benefit from continued treatment in the opinion of the parent study investigator from dosing of TJ004309 in combination with atezolizumab.
2. Willing or able to comply with study treatment and standard of care testing and procedures.

Exclusion Criteria:

1. Any unresolved ongoing toxicity or clinical event that would make continued treatment with TJ004309 inappropriate.
2. Current treatment in another clinical study or treatment with other standard of care therapy.
3. Currently pregnant.
4. Current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might interfere with the patient's participation or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Arizona Oncology Associates, P.C., Tucson, Arizona